CLINICAL TRIAL: NCT07222111
Title: Prebiotics in Women's Health and Aging: The Gut-Bone Connection
Brief Title: Prebiotics (Dried Plum) and Immune Function in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other); Purdue University (Other)
Responsible Party: Principal Investigator, Brenda J. Smith, Professor and Vice-chair of Translational Research in OBGYN, Indiana University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB# 23232; 2024-67017-42495 (Other Grant/Funding Number: USDA-NIFA)
Record Dates: First submitted 2025-09-01; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: T Cell Response to Dried Plum; Vitamin D Influence on Immune Response; Dried Plum and Immune Function
Keywords: immune system; dried plums; prebiotics; T cells; bone health; vitamin D

STUDY DESIGN:
Intervention Model Description: The two study arms are normal diet (control) or normal diet supplemented with dried plum (intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dried Plum (Experimental): Participants will consume their usual diet supplemented with 50 g of dried plum (5-6 dried plums) per day.
  Interventions: Dietary Supplement: Dried plums
- Regular Diet (No Intervention): Participants will consume their usual diet.

INTERVENTIONS:
Dietary Supplement: Dried plums — Participants will supplement their regular diet with 50 g of dried plum (5-6 dried plums) per day.
  Arms: Dried Plum

SUMMARY:
Prior studies have shown that dietary supplementation with dried plums (also known as prunes) reduces bone loss in postmenopausal women. The purpose of this clinical trial is to understand how dried plums mediate their effects on bone. The main questions the study will answer are:

1. Does adding dried plums to the diet alter immune cell function?
2. Does dried plum alter gut microbes?
3. Does a person's vitamin D status influence this response?

Researcher will compare the response following consumption of the normal diet to supplementing the diet with dried plums.

Participant will:

1. Consume their normal diet or supplement their normal diet dried plums for four week periods over the course of 3-4 months.
2. Complete 5 study visits scheduled.
3. Perform some physical function tests and have a bone density scan at the beginning of the study.
4. Complete questionnaires, a 3-day food record, and provide stool and blood samples at 4 different timepoints during the study.
5. Record information about their bowel habits

DETAILED DESCRIPTION:
Each year in the U.S., an estimated 2 million women (~6,000 women each day) reach the critical stage of female reproductive aging known as menopause. Menopause is characterized by the permanent cessation of menses and the loss of ovarian follicular activity brought about by the decline in 17β-estradiol (i.e., estrogen deficiency). Among American women, the median age of menopause is 51 y [1]. Based on a current life expectancy of 80.5 yrs, women in this country can expect to spend up to one-third of their lifetime in this postmenopausal stage.

The impact of decreasing 17β-estradiol on immune cell function, especially some T cell populations, has become the focus of much women's health research. It is widely accepted that after menopause women exhibit a significant increase in their risk for chronic diseases, including gynecologic and breast cancers, autoimmune diseases, cardiovascular disease, and osteoporosis. In terms of bone health, which is the focus of our laboratory's work, postmenopausal women are 4 times more likely to fracture compared to pre-menopausal women (age 20-50 yrs). Moreover, 1 in 3 women over the age of 50 y will experience an osteoporotic fracture. The decline in 17β-estradiol that occurs with menopause is accompanied by immunological changes in cluster of differntiation (CD)4+ effector T cells, most notably an increase in T helper cells expressing the pro-inflammatory cytokine, interleukin (IL)-17 (i.e., Th17 cells) relative to the immunosuppressive, T regulatory (Treg) cells. Th17 cells are highly potent promoters of osteoclastogenesis and accelerate the bone resorption that occurs in estrogen deficiency. In contrast, the osteoprotective role of Tregs, which are reported to either decrease or remain unchanged in with menopause, is less clear in humans beyond their anti-inflammatory properties. Consequently, it is the increase in Th17 cells that is the major determinant of the altered Treg/ Th17 ratio that is reported in response to declining estrogen and has a central role in the pathophysiology of postmenopausal osteoporosis.

Recent evidence has revealed that the gut microbiota is a critical regulator of this osteoimmunological (i.e., T cell) response; thus, establishing the gut-bone axis as a viable target to prevent estrogen deficiency-induced bone loss. Clinical studies have shown that utilizing probiotics and prebiotics to alter the gut microbiota has beneficial effects on bone and mineral metabolism. In animal models of postmenopausal osteoporosis, probiotics and prebiotics increase gut-derived metabolites (e.g., short chain fatty acids (SCFA)), program more tolerogenic or anti-inflammatory immune responses, while preventing bone loss. Our laboratory's extensive work on dried plum and its unique ability to not only prevent, but also reverse bone loss in animal models, has revealed that it improves T cell function ex vivo and both its polyphenolic and carbohydrate components contribute to its prebiotic activity. These findings combined with strong evidence from three separate clinical trials support the ability of dried plum to prevent postmenopausal bone loss [1-3] make it an excellent prebiotic candidate to test whether these gut-mediated changes in immune function observed in animal models translate to human subjects.

In addition to age-related changes in estrogen, other factors affecting the T cell biology of postmenopausal women (e.g., vitamin D status) could further compound their osteoporosis risk. Among U.S. women age 51-70 yrs, 28% are vitamin D insufficient and 10% are vitamin D deficient based on the Institute of Medicine guidelines. Although vitamin D is known for its role in skeletal health, evidence of its important extraskeletal functions continues to emerge. 1,25-(OH)2D3 simultaneously inhibits the pro-inflammatory Th17 cell and increases the anti-inflammatory Treg cell, number and function. Furthermore, vitamin D's influence on immune function has been recently linked, albeit indirectly, to the gut microbiota. Thus, postmenopausal women who have compromised vitamin D status may face even greater risk of T cell-mediated pathologies (e.g., autoimmune diseases & osteoporosis), which further highlights the importance of targeting the gut microbiota.

The goal of this study is to understand how dietary supplementation with dried plums, a food with prebiotic activity, affects T effector cells (i.e., Th17 & Treg) and their function; and to explore whether vitamin D status of the host alters this response. The fundamental questions to be addressed are: 1) whether supplementing the diet with dried plum affects immune function (i.e., T effector cells); 2) whether the findings of our pre-clinical studies demonstrating the gut microbiota is a target to counter T cell changes associated with estrogen deficiency translate to postmenopausal women; and 3) whether the vitamin D status of the host influences the response to this prebiotic.

To accomplish this, we will recruit healthy postmenopausal women, age 60-75 years, to participate in a randomized crossover control trial with and without dried plum. We plan to enroll n=30 women. Eligible volunteers will complete 5 study visits at the Clinical Research Center at the IU Health University Hospital. At Visit 1, volunteers will undergo screening to ensure they are eligible to participate and after giving informed consent, they will have anthropometrics, a baseline bone density scan and physical function assessments. Prior to Visit 2, and all subsequent visits, participants will collect stool samples and enter their 3-day diet record into the Automated Self-administered 24-hour (ASA24).

The primary study visits (Visits 2-5) are divided into two arms (each 4 wks in duration with 1 wk run-in) and a washout period (2-4 wks). At Visit 2, participants will then be randomly assigned to the Arm A (with dried plum intervention) or Arm B (without the dried plum intervention) using a computer-generated list of random numbers. When participants are on Arm A, instructions will be provided on the run-in protocol and incorporating dried plum into the diet (50 g/day or 5-6 dried plums per day). Participants will record the amount and time of day the dried plums are consumed and return any remaining product. Study personnel will provide the dried plums in snack packs at no cost. Note the snack packs are provided by the California Prune Board. At Visit 3, participants will complete the data and sample collection as described for Visit 2 and then begin the washout period. Visit 4 will be scheduled following the washout period and the same procedures described in Visit 3 will be repeated with crossover to the second arm. At Visit 5 (final visit), participants will complete the data and sample collection.

At Visits 2-5, participants will also complete physical activity and sun exposure questionnaires. They will provide a blood sample, and update study personnel about any changes in their health status. Throughout both arms of the study, participants will rate their bowel habits on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* women 60-75 years of age at the start of the study;
* 12 or more consecutive months without a menstrual period;
* willing to include dried plums in their daily diet and collect fecal samples at four time points;
* ambulatory without assistance;
* capacity to give informed consent.

Exclusion Criteria:

* women who have been on medications known to alter bone or calcium metabolism (e.g., oral bisphosphonates, raloxifene, denosumab, intermittent parathyroid hormone, growth hormone) within 12 months of starting the study. Prior use of intravenous bisphosphonates at any time.
* women who have been on hormone replacement therapy, steroids (i.e., glucocorticoids), biologics, or chronic NSAID within 3 months of starting the study.
* women with a previous diagnosis of osteoporosis (i.e., BMD T-score or history of vertebral fracture or fragility fractures of hip, wrist, humerus after the age of 50 yr) or other metabolic bone disease (e.g., osteomalacia or osteogenesis imperfect), renal disease, stroke, heart attack, type 2 diabetes, liver disease or autoimmune diseases (e.g., rheumatoid arthritis, systemic Lupus erythematosus, type 1 diabetes mellitus, IBD) that could affect bone metabolism or T cell biology will be excluded.
* women who have undergone treatment for cancer within 12 months of starting the study
* women who have been taking prebiotic or probiotic supplements or natural products that have estrogen-like effects in the past 3 months
* women who smoke, have a BMI >40 kg/m2 or <18.5 kg/m2, or consume >2 alcoholic drinks per day
* women who regularly consume dried plums or prune juice (>1 serving weekly).

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Circulating T Helper (Th)17 Cells | Change from baseline to the end of each 4-week arm of the study
  Change in the relative abundance of circulating Th17 cells in response to dried plum supplementation compared to control arm of the study will be reported.
Ex Vivo T Cell Function | The end of each 4 week arm of the study
  Ex vivo experiements will be performed with peripheral blood mononuclear cells (PBMCs) collected at the final time points of each of the two arms (4 weeks in duration) of the study. Cells will be challenged and the release of interleukin 17 and interleukin 10 will be assessed in the media. The cytokine response of cells collected at the end of the control or dried plum treatment arm arm will be assessed.
Treatment Effects on Serum IL-6 | End of the 4-week control and dried plum treatment arm of the study.
  Serum IL-6 will be compared at the end of the control arm and at the end of dried plum supplementation arm of the study.

SECONDARY OUTCOMES:
Change in Circulating T Regulatory Cells | Change from baseline to the end of each 4-week arm of the study
  The change in the relative abundance of circulating T regulatory (Treg) cells in response to dried plum supplementation compared to control arm of the study will be reported .
Change in the Treg to Th17 ratio | The change from baseline until final time points of each arm of each 4-week arm of the study.
  The change in the relative abundance of Treg and Th17 cells (as previously described) will be expressed as a ratio to determine if the Treg:Th17 cell ratio is altered in response to treatment with dried plum.
Ex Vivo T Cell TNF-a | Sample collected at the end of each 4-week arm of the study
  Ex vivo experiements will be performed with peripheral blood mononuclear cells (PBMCs) collected at the final time points of each of the two arms (4 weeks in duration) of the study. Cells will be challenged and the release of tumor necrosis factor-alpha (TNF-a) will be assessed in the media. The cytokine response of cells collected at the end of the control or dried plum treatment arm arm will be assessed.
Change in Serum Metabolites | The change from baseline until final time points of each arm of each 4-week arm of the study.
  The change in the abundance of serum metabolites will be assessed in response to treatment arm with dried plum compared to the control arm of the study.
Change in Fecal Metabolites | The change from baseline until final time points of each arm of each 4-week arm of the study.
  The change in the abundance of fecal metabolites will be assessed in response to the treatment arm with dried plum compared to the control arm of the study.
Change in Fecal Microbiota | The change from baseline until final time points of each arm of each 4-week arm of the study.
  Change in the fecal microbiota profile will be evaluated bewteen baseline and final time points of the treatment arm (with dried plum) and the control arm of the study.
Serum Pro- and Anti-inflammatory Cytokines | End of the 4-week control arm and 4-week dried plum arm of the study.
  Differences between serum tumor necrosis factor alpha (TNF-a) and interleukin IL-10 will be compared at the end of the control arm and at the end of dried plum supplementation arm of the study.
Serum C-telopeptide I (CTX-1) | Time Frame: End of the 4-week control arm and 4-week dried plum arm of the study.
  Serum C-telopeptide I (CTX-1), a biomarker of bone resorption, will be assessed at the end of the control arm and at the end of dried plum supplementation arm of the study.

OTHER OUTCOMES:
Dietary Assessment | Baseline and at the completion of each 4-week arm of the study.
  Participants will complete a 3-day food record using the ASA24 pre- and post- each arm of the study. Dietary assessment include at a minimum kcal intake and macronutrient composition.
Physical Activity Assessment | Prior to and at the completion of each 4-week arm of the study
  Using the CHAMPS Physical Activity for Older Adults Questionnaire will be completed pre- and post- each arm of the study. The information will be used to characterize usual activity level and consistency during the study.
Body weight | Prior to and at the completion of each 4-week study arm
  Weight will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health University Hospital Clinical Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
As described above, the compiled data will be kept in the IU's institutional repository, IU ScholarWorks. Deposition of (de-identified) data in this system creates a DOI that will be used in publications to facilitate discovery. We will share metadata as well as participant data associated with the study. Data will be made available to investigators with PD permission and consistent with the USDA and the university guidelines. Data will be deposited in the IU ScholarWorks and embargoed for one year after the completion of the study. We will provide the names and institutions of persons who were either given or denied access to the data, and the bases for such decisions will be included in the annual progress report.
Supporting Information: Study Protocol
Time Frame: August 2029
Access Criteria: Investigators with PI permission

REFERENCES:
- [Background] Hooshmand S, Kern M, Metti D, Shamloufard P, Chai SC, Johnson SA, Payton ME, Arjmandi BH. The effect of two doses of dried plum on bone density and bone biomarkers in osteopenic postmenopausal women: a randomized, controlled trial. Osteoporos Int. 2016 Jul;27(7):2271-2279. doi: 10.1007/s00198-016-3524-8. Epub 2016 Feb 22. PMID 26902092
- [Background] Hooshmand S, Chai SC, Saadat RL, Payton ME, Brummel-Smith K, Arjmandi BH. Comparative effects of dried plum and dried apple on bone in postmenopausal women. Br J Nutr. 2011 Sep;106(6):923-30. doi: 10.1017/S000711451100119X. Epub 2011 May 31. PMID 21736808
- [Background] De Souza MJ, Strock NCA, Williams NI, Lee H, Koltun KJ, Rogers C, Ferruzzi MG, Nakatsu CH, Weaver C. Prunes preserve hip bone mineral density in a 12-month randomized controlled trial in postmenopausal women: the Prune Study. Am J Clin Nutr. 2022 Oct 6;116(4):897-910. doi: 10.1093/ajcn/nqac189. PMID 35798020
- See also: All IN for Health is a platform made availabe through the NIH supported, Indiana Clinical and Translational Sciences Institute to improve resident's participation in clinical trials. — https://research-studies.allinforhealth.info/us/en/listing/13151/prebiotics-in-womens-health/?&nctidentifier=tx13151

DOCUMENTS (2):
  • Study Protocol (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT07222111/Prot_000.pdf
  • Informed Consent Form (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT07222111/ICF_001.pdf